CLINICAL TRIAL: NCT05121597
Title: Nasotracheal Intubation in Dental Treatments Under General Anesthesia in Children: Comparison of Direct Macintosh Laryngoscopy and HugeMed Video Laryngoscopy
Brief Title: The Comparison of Direct Macintosh Laryngoscopy and HugeMed Video Laryngoscope for Nasotracheal Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ozlem Kocaturk, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OKocaturk
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Intubation; Difficult or Failed; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscope Group (Experimental): The group that we will use a videolaryngoscope for nasotracheal intubation.
  Interventions: Device: HugeMed Videolaryngoscope
- Control Group (Active Comparator): The group that we will use a direct laryngoscope for nasotracheal intubation.
  Interventions: Device: HugeMed Videolaryngoscope

INTERVENTIONS:
Device: HugeMed Videolaryngoscope — Macintosh laryngoscope
  Other Names: Direct laryngoscope

SUMMARY:
Forty-four patients aged 4-10 years who applied to Aydın Adnan Menderes University Faculty of Dentistry for dental treatment under general anesthesia will be selected and divided into 2 groups by simple randomization. The group in which a direct laryngoscope was used for intubation, which is a part of the routine general anesthesia procedure, Group DL; The group in which the video laryngoscope is used will be called Group VL. Routine general anesthesia procedure and dental treatments will not differ between groups. The necessity of external laryngeal manipulation, intubation difficulty scale (IDS) will be evaluated and the difficulty level will be determined as easy, medium and difficult. All intubations will be confirmed by auscultation as part of the routine procedure.

DETAILED DESCRIPTION:
Forty-four patients aged 4-10 years who applied to Aydın Adnan Menderes University Faculty of Dentistry for dental treatment under general anesthesia will be included and divided into 2 groups randomly. The group in which a direct laryngoscope was used for intubation, which is a part of the routine general anesthesia procedure, Group DL; The group in which the video laryngoscope is used will be called Group VL.

Routine general anesthesia procedure and dental treatments will not differ between groups. The time from the moment the laryngoscope touches the patient until the endotracheal tube is inserted and the end-tidal carbon dioxide is detected will be recorded as intubation time, and the Cormack and Lehane glottic scale score will be recorded when the best glottic view is obtained. The necessity of external laryngeal manipulation, intubation difficulty scale (IDS) will be evaluated and the difficulty level will be determined as easy, medium and difficult. All intubations will be confirmed by auscultation as part of the routine procedure.

Desaturation (SpO2 < 90%) will be assessed during intubation, Hemodynamic data will be recorded at four points in time: at baseline (before induction, T0); 1 min after induction (T1); in intubation (T2); and 5 minutes after intubation (T3).

Intubation time, Intubation Difficulty Scale (IDS), C&L grade, number of intubation attempts, External Throat Manuplation, Intubation related trauma-bleeding, Intubation-related pain scores will be recorded in the case report form. In addition, age, gender, weight, ASA status of patients, blade and tube size, operation time, number of caries-filled extracted teeth (dmft) values will also be recorded. The patient whose operation is completed will be taken to the recovery room. Post-operative discomfort will be recorded in the case report form.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-10 years who cannot undergo dental treatment in a routine clinical setting (having a Frankl 1 and 2 behavior score) due to lack of cooperation,
* ASA (American Society of Anesthesiologist) Score 1 (no systemic disease),
* Cases with Mallampati Score I-II.

Exclusion Criteria:

* Suspect or history of difficult intubation,
* BMI (body mass index) greater than 35,
* Fast-series induction required,
* Nasal intubation is contraindicated,
* Cases in which general anesthesia is contraindicated (Drug allergies, advanced systemic disease, muscle diseases, etc.)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Intubation difficulty scale | At the time of intubation
  Difficulty level of intubation will be determined as easy, medium and difficult.
  The 3 classifications were as follows: if the IDS was 0 points, then it was considered an easy endotracheal intubation. If the score was 1-5 points, it was a slightly difficult intubation. More than 5 points was considered moderate-to-difficult intubation.

SECONDARY OUTCOMES:
Postoperative throat pain | Postoperative 1 hour
  Postoperative pain due to intubation was evaluated by visual analogue scale (VAS).
  Pain visual analog scale (VAS) score (0-10, 0 indicating no pain, 10 indicating the intolerable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We wiil not share individual participant data (IPD).

REFERENCES:
- [Background] Kim EH, Lee JH, Song IK, Kim JT, Kim BR, Kim HS. Effect of head position on laryngeal visualisation with the McGrath MAC videolaryngoscope in paediatric patients: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jul;33(7):528-34. doi: 10.1097/EJA.0000000000000448. PMID 26986776
- [Derived] Kocaturk O, Keles S. Comparison of the HugeMed video laryngoscope with the Macintosh direct laryngoscope for nasotracheal tracheal intubation in children undergoing dental treatment: a randomized controlled clinical study. Expert Rev Med Devices. 2024 Jun 3:1-8. doi: 10.1080/17434440.2024.2363289. Online ahead of print. PMID 38829609